CLINICAL TRIAL: NCT06989177
Title: An Interventional Study Investigating the Effects of Probiotics on Body Weight and Metabolic Homeostasis
Brief Title: Probiotic Intervention on Body Weight
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIAS-PITBW-202503
Record Dates: First submitted 2025-05-06; First posted 2025-05-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Homeostasis; Weight Loss; Probiotic Intervention
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Probiotics; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (Placebo Comparator): They will receive energy-restricted nutritional and lifestyle intervention and placebo
  Interventions: Behavioral: Energy-restricted nutritional and lifestyle intervention; Dietary Supplement: Placebo
- GLP-1RA Group (Active Comparator): They will receive an energy-restricted nutritional and lifestyle intervention , in conjunction with prescribed semaglutide therapy.
  Interventions: Behavioral: Energy-restricted nutritional and lifestyle intervention; Drug: semaglutide
- Probiotic Group (Experimental): They will receive an energy-restricted nutritional and lifestyle intervention and LC-19
  Interventions: Behavioral: Energy-restricted nutritional and lifestyle intervention; Dietary Supplement: Probiotic
- Healthy Comparators (Other): They will receive general lifestyle and nutritional education.
  Interventions: Behavioral: General lifestyle and nutritional education

INTERVENTIONS:
Behavioral: General lifestyle and nutritional education — Participants will receive dietary advice, behavior guidance and nutritional and lifestyle education based on dietary guidelines.
  Arms: Healthy Comparators
Behavioral: Energy-restricted nutritional and lifestyle intervention — Participants will receive dietary advice, behavioral guidance and nutritional and lifestyle education by dietitian and physicians. App-connected wearable devices will be utilized to monitor their dietary intakes and App-connected scale will be used to monitor their weight changes during interventions.
  Arms: Control Group; GLP-1RA Group; Probiotic Group
Dietary Supplement: Placebo — Participants will receive one bag (2 g; 1 × 10¹² CFU) daily of LC-19.
  Arms: Control Group
Dietary Supplement: Probiotic — participants will receive daily one bag of LC-19 (10^12 cfu/bag).
  Arms: Probiotic Group
Drug: semaglutide — Participants will receive prescibed semaglutide therapy
  Arms: GLP-1RA Group

SUMMARY:
This study is a randomized controlled trial with 120 overweight or obese (body-mass index, BMI, ≥ 24 kg/m²) participants and 20 normal-weight participants. Twelve weeks of energy-restricted nutritional and lifestyle intervention with placebo, Lactobacillus paracasei LC-19 (LC-19), or semaglutide (a glucagon-like peptide-1 receptor agonist, GLP-1RA) will be randomly conducted in the overweight or obese participants. The primary goal is to clarify the roles of LC-19 and semaglutide in weight reduction and in improving energy, glucose, and lipid metabolism, while also comparing side effects, adverse events, and long-term outcomes such as weight regain between these two interventions. In addition, the study will explore key factors affecting intervention response to provide evidence for optimizing individualized intervention strategies.

DETAILED DESCRIPTION:
The primary goal is to clarify the roles of LC-19 and semaglutide in weight reduction and in improving energy, glucose, and lipid metabolism, while also comparing side effects, adverse events, and long-term outcomes such as weight regain between these two interventions. In addition, the study will explore key factors affecting intervention response to provide evidence for optimizing individualized intervention strategies.

In this study, 120 overweight or obese participants (BMI ≥ 24 kg/m²) will be recruited and be randomly assigned to one of the three groups: an energy-restricted nutritional and lifestyle intervention + placebo group (control group), an energy-restricted nutritional and lifestyle intervention plus LC-19 group (probiotic group), or an energy-restricted nutritional and lifestyle intervention plus semaglutide injection group (GLP-1RA group), with a 12-week intervention. In addition, 20 normal-weight participants will be recruited and receive 12-week weight maintenance nutritional and lifestyle interventions. Before and after the 12-week interventions, metabolic homeostasis will be used to characterize metabolic health and to be determined using comprehensive measurements of dynamic changes in postprandial metabolic responses (including energy metabolism, multiple clinical biomarkers, metabolomic signatures, gut microbiota, genetic signatures etc.) after the standardized mixed-meal tolerance test (MMTT; 126.5 g glucose, 30.67 g fat and 34.5 g protein) in whole-room indirect calorimeter under resting conditions. In addition, data from dietary intake, anthropometric measurements, body composition, behavior questionnaires, 14-day continuous glucose monitoring, and 14-day accelerometer-based physical activity and sleep monitoring will also be collected to characterize metabolic homeostasis. During the interventions, participants will receive dietary advice, behavior guidance and nutritional and lifestyle education by dietitian and physicians. App-connected wearable devices will be utilized to monitor their dietary intakes and an app-connected scale will be used to monitor their weight changes during interventions. Additionally, at 6 months post-intervention, a follow-up assessment will be conducted, including questionnaires (consistent with the baseline visit), anthropometry (e.g., height, weight, waist and hip circumference, blood pressure, pulse), clinical laboratory tests (e.g., blood glucose, blood lipids, liver and kidney function), and stool sample collection. The study protocol has been approved by the Ethics Committee of Tongde Hospital of Zhejiang Province.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 50 years.
* Normal-weight participants: 18.5 kg/m² ≤ Body Mass Index (BMI) < 24 kg/m².
* Overweight or obese participants:

BMI ≥ 28 kg/m², or 24 kg/m² ≤ BMI < 28 kg/m² and a clinical diagnosis meeting semaglutide treatment indications (e.g., hyperglycemia, hypertension, dyslipidemia, fatty liver, obstructive sleep apnea, cardiovascular disease, etc.).

* Willingness to participate in this study and provide signed informed consent.

Exclusion Criteria:

* Abnormal metabolic indicators (meeting any one of the following criteria is grounds for exclusion):

  1. Normal weight (18.5 kg/m² ≤ BMI < 24 kg/m²):
  1. Waist circumference ≥ 90 cm for men or ≥ 85 cm for women.
  2. Fasting glucose ≥ 6.1 mmol/L or 2-hour postprandial glucose ≥ 7.8 mmol/L, or a confirmed diagnosis of diabetes.
  3. Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg, or currently under antihypertensive treatment.
  4. Fasting triglycerides (TG) ≥ 1.7 mmol/L; high-density lipoprotein cholesterol (HDL-C) < 0.9 mmol/L in men or < 1.0 mmol/L in women.

  2. Overweight or obese (BMI ≥ 24 kg/m²):
  1. Fasting plasma glucose > 11.1 mmol/L or HbA1c > 9%, or previously diagnosed diabetes, or currently using insulin or any antidiabetic medication.
  2. Blood pressure ≥ 160/100 mmHg, or clinically diagnosed stage 2 or stage 3 (moderate or severe) hypertension, or currently under antihypertensive treatment.
  3. Use of lipid-lowering drugs (e.g., fibrates, bile acid sequestrants, statins, PCSK9 inhibitors) within the past 3 months, or TG ≥ 5.7 mmol/L, or LDL ≥ 4.9 mmol/L.
* Pregnancy or lactation.
* Self-reported weight change of more than 5 kg within the 90 days prior to screening.
* Use of antibiotics, antimicrobials, or anti-inflammatory/analgesic salicylates (e.g., aspirin) within the 3 months prior to screening for 3 days or more.
* Use of estrogen therapy or other hormonal medications within the past 6 months.
* Use of GLP-1 receptor agonists or probiotics within the past 3 months.
* Heavy alcohol consumption (females > 40 g/day, approximately 250 mL of huangjiu [yellow rice wine], or 1000 mL of beer, or 100 mL of liquor per day; males > 80 g/day).
* Severe liver or kidney dysfunction (ALT, AST, or serum creatinine exceeding 3 times the upper limit of normal, UACR ≥ 30 mg/g, or eGFR < 60 mL/min).
* Gastrointestinal diseases affecting digestion and absorption (e.g., severe diarrhea, severe constipation, severe inflammatory bowel disease, peptic ulcer, gallstones, cholecystitis).
* Underwent surgery within the past year (excluding appendectomy or hernia repair).
* Severe cardiovascular or cerebrovascular diseases (e.g., heart failure, myocardial infarction, stroke, acute myocarditis, severe arrhythmia, or receiving interventional therapy).
* Presence of metallic implants such as a cardiac stent or pacemaker.
* Cancer or having received radiation or chemotherapy within the past 5 years.
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia, or a personal history of hyperthyroidism or hypothyroidism.
* Chronic or acute pancreatitis.
* Positive hepatitis B surface antigen (HBsAg), active tuberculosis, HIV, or other infectious diseases.
* Currently participating in another clinical study or having done so within the past 3 months.
* Claustrophobia.
* Any psychiatric disorder such as attention-deficit/hyperactivity disorder (ADHD), bipolar disorder, or epilepsy (including current use of antiepileptic medications), or use of antidepressant medications.
* Inability to read, write, operate a smartphone, or perform daily activities independently.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight (kg) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Weight will be assessed using a Seca 255 scale (ScalesGalore).

SECONDARY OUTCOMES:
Change in Energy Expenditure Rate (kcal/min) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Energy expenditure rate (kcal/min) will be assessed with a whole-room indirect calorimeter (Sable).
Change in Respiratory Quotient from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Respiratory quotient will be assessed with a whole-room indirect calorimeter.
Change in Fat Oxidation Rate (g/min) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Fat oxidation rate (g/min) will be assessed with a whole-room indirect calorimeter.
Change in Carbohydrate Oxidation Rate (g/min) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Carbohydrate oxidation rate (g/min) will be assessed with a whole-room indirect calorimeter.
Change in Waist Circumference (cm) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Waist circumference will be assessed with a Seca 201 tape (ScalesGalore).
Change in Hip Circumference (cm) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Hip circumference will be assessed with a Seca-201 tape (ScalesGalore).
Change in Fat Mass (kg) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Fat mass will be assessed using dual energy x-ray absorptiometry (DXA; GE).
Change in Fat-free Mass (kg) from Baseline to Week 12 | Baseline (week 0) and Week 12
  The change from baseline to after the 12-week intervention. Fat-free mass will be assessed using DXA (GE).
Change in Controlled Attenuation Parameter (CAP, dB/m) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. CAP will be assessed using FibroScane (Echosens). The median CAP value of 10 valid measurements will be used (IQR ≤ 30%). Reported value = Week 12 CAP minus baseline CAP; positive values indicate increased hepatic steatosis.
Change in Systolic Blood Pressure (mmHg) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Systolic blood pressure will be assessed with an Omron J750 electronic monitor.
Change in Diastolic Blood Pressure (mmHg) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Diastolic blood pressure will be assessed with an Omron J750 electronic monitor.
Change in Heart Rate (beats/min) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Heart rate will be assessed with an Omron J750 electronic monitor.
Change in Fasting Glucose (mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Glucose will be measured using a hexokinase enzymatic assay.
Change in Glucose Incremental AUC (mmol·min/L) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an oral mixed-meal tolerance test (MMTT). Glucose will be measured using a hexokinase enzymatic assay. Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in HbA1c (%) from Baseline to Week 12 | Baseline (Week 0) and Week 12
  The change from baseline to after the 12-week intervention. HbA1c will be assessed using high-performance liquid chromatography.
Change in Mean 24-h Glucose (mg/dL) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Mean 24-h glucose will be assessed using Continuous Glucose Monitoring (FreeStyle Libre 2, Abbott) for 14 consecutive days.
Change in Glucose Coefficient of Variation (CV, %) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Glucose CV will be calculated as (SD / mean) × 100% from continuous glucose monitoring (FreeStyle Libre 2, Abbott) over 14 consecutive days.
Change in Fasting Insulin (µIU/mL) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Insuin will be measured using an electrochemiluminescence assay.
Change in Insulin Incremental AUC (µIU·min/mL) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. Insulin will be measured using an electrochemiluminescence assay. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Fasting C-peptide (ng/mL) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. C-peptide will be measured using an electrochemiluminescence assay.
Change in C-peptide Incremental AUC (ng·min/mL) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. C-peptide will be measured using an electrochemiluminescence assay. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Fasting Serum Triglycerides (mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Serum triglycerides will be quantified using an enzymatic colorimetric assay.
Change in Triglyceride Incremental AUC (mmol·min/L) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. Triglyceride will be measured using an enzymatic colorimetric assay. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Serum Fasting Total Cholesterol (mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. Total cholesterol will be quantified in serum using an enzymatic colorimetric assay.
Change in Total Cholesterol Incremental AUC (mmol·min/L) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. Total cholesterol will be measured using an enzymatic colorimetric assay. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Fasting Serum High-Density Lipoprotein Cholesterol (HDL-C, mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. HDL-C will be quantified in serum using an enzymatic colorimetric assay.
Change in HDL-c Incremental AUC (mmol·min/L) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. HDL-c will be measured using an enzymatic colorimetric assay. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Fasting Serum Low-Density Lipoprotein Cholesterol (LDL-C, mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change from baseline to after the 12-week intervention. LDL-C will be quantified in serum using an enzymatic colorimetric assay.
Change in LDL-c Incremental AUC (mmol·min/L) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240 and 300 min during an MMTT. LDL-c will be measured using an enzymatic colorimetric assay. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in GLP-1 Incremental AUC (pg·min/mL) from Baseline to Week 12 | Baseline (Week 0) and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240 and 300 min during an MMTT. GLP-1 will be quantified using a high-sensitivity ELISA. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value.
Change in GIP Incremental AUC (pg·min/mL) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. GIP will be quantified using a high-sensitivity ELISA. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value.
Change in Ghrelin Incremental AUC (pg·min/mL) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. Ghrelin will be quantified using a high-sensitivity ELISA. iAUC will be calculated via the trapezoidal rule after subtracting the fasting value.
Change in Shannon Diversity Index from Baseline to Week 12 | Baseline and Week 12
  Fecal DNA will be extracted and subjected to shotgun metagenomic sequencing on an Illumina NovaSeq 6000 (2 × 150 bp; ≥6 Gb per sample). Reads will be taxonomically profiled using MetaPhlAn 4.0. The Shannon diversity index will be calculated for each sample. Reported value = Week 12 index - baseline index.
Change in Relative Abundance of Akkermansia muciniphila (%) from Baseline to Week 12 | Baseline and Week 12
  Same sequencing workflow as above. Relative abundance (% of total classified reads) of A. muciniphila will be extracted from MetaPhlAn output. Reported value = Week 12 abundance - baseline abundance.
Single Nucleotide Polymorphisms (SNPs) | Baseline
  Mutations at specific sites will be detected using a genotyping microarray.
Change in body weight from Week 12 to 6 months post-intervention | Post-intervention 6 months
  The change from the end of intervention (Week 12) to 6 months post-intervention. Weight will be assessed using a Seca-255 scale (ScalesGalore).

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Institute for Nutritional Sciecnes, CAS; Hangzhou Institute for Advanced Study, UCAS
Locations (1):
- Hangzhou Institute for Advanced Study, University of Chinese Academy of Sciences, Hangzhou, Zhejiang, China